CLINICAL TRIAL: NCT02557438
Title: Bone Metabolism in Adolescents Undergoing Bariatric Surgery
Brief Title: Effects of Weight Loss Surgery on Bone Health in Adolescents
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Madhusmita Misra, Professor of Pediatrics, Massachusetts General Hospital
Other Study IDs: 2015P000360
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Surgery
Keywords: Bone; Child Health; Nutrition
MeSH Terms: conditions — Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, fecal samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Roux-en-Y Gastric Bypass: Males and females aged 13-25 undergoing Roux-en-Y gastric bypass (RYGB) surgery
  Interventions: Procedure: Roux-en-Y Gastric Bypass
- Vertical Sleeve Gastrectomy: Males and females aged 13-25 undergoing vertical sleeve gastrectomy (VSG) surgery
  Interventions: Procedure: Vertical Sleeve Gastrectomy
- Non-surgical Obese Controls: Males and females aged 13-25 who are obese and not undergoing weight loss surgery

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass — Determination of the kind of surgery will be made by the participant's providers and not by study staff
  Other Names: RYGB
  Groups: Roux-en-Y Gastric Bypass
Procedure: Vertical Sleeve Gastrectomy — Determination of the kind of surgery will be made by the participant's providers and not by study staff
  Other Names: VSG
  Groups: Vertical Sleeve Gastrectomy

SUMMARY:
The purpose of this study is to examine the impact of weight-loss surgery (Roux-en-Y gastric bypass or Vertical Sleeve Gastrectomy) on bone outcomes in girls and boys ages 13-21. This study will also examine a group of overweight boys and girls who are not scheduled or planned for surgery for comparison of these outcomes.

Obese adults who undergo weight-loss surgery are at risk for bone loss and decreased bone strength. The investigators do not know the effects of such surgery on bone in teenagers and young adults. The purpose of this study is to find out how different types of weight loss surgery affect bone density and strength in teenagers and young adults and compare these results to obese teenagers and young adults who are not undergoing weight-loss surgery.

DETAILED DESCRIPTION:
Our overall hypothesis is that both Roux-en-Y Gastric Bypass (RYGB) and vertical sleeve gastrectomy (VSG) in adolescents with morbid obesity will lead to a reduction in areal and volumetric BMD, and deterioration in bone structure and estimated bone strength, and an increase in marrow adiposity. We further hypothesize that these effects will be due in part to a decrease in lean mass, changes in enteric peptide hormones and reduced estrogen levels.

We will enroll 120 participants 13-21 years old for this two-year longitudinal study (36 in each of the surgical groups and 48 non-surgical controls with obesity). We will screen up to 240 subjects to find these 120 eligibile subjects. Areal bone mineral density (BMD) will be assessed by dual energy x-ray absorptiometry (DXA), volumetric BMD by quantitative computed tomography (QCT), bone structure and strength using high resolution peripheral QCT and finite element analysis, and marrow fat using magnetic resonance spectroscopy. Body composition will also be assessed.

Adolescence is a critical time for bone accrual and the use of bariatric procedures is increasing in teenagers. This study will provide novel data needed to establish effects of RYGB vs. VSG on bone in adolescents and will begin to delineate underlying mechanisms. Clarifying these mechanisms will identify therapeutic targets to optimize bone accrual in adolescents undergoing bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents with morbid obesity 13-25yo undergoing RYGB (n=36) or VSG (n=36), or being followed without surgical intervention (usual care) (n=48).
2. Eligibility criteria for weight loss surgery used at the Weight Center include BMI>40 or BMI>35kg/m2 with major comorbidities. A BMI>35 in adolescents reflects a BMI>99th percentile. In order to be considered appropriate surgical candidates, children must have a bone age of ≥14y (F) or ≥16y (M), and ≥1 co-morbidity of obesity. They must have demonstrated efforts at non-surgical weight loss, and consistent compliance with appointments and recommendations. Patients must demonstrate sufficient maturity, psychological stability and cognitive capacity to recognize the significance of the procedure and implement required post-operative behavioral changes.

Exclusion Criteria:

1. Current pregnancy and breast feeding
2. Medications other than calcium or vitamin D that affect bone, such as glucocorticoids, phenytoin, phenobarbitone (washout of 3 months prior to enrollment if discontinuation is medically permissible)
3. Use of antipsychotic medications that cause weight gain if treated for <6 mos, or if dosage is not stable for >2 mos
4. Untreated thyroid dysfunction or on stable dose for <3 mos
5. HbA1C>8% (to avoid deleterious effects on bone from uncontrolled T2DM)
6. Smoking >10 cigarettes/day; substance abuse per Diagnostic and Statistical Manual (DSM) V
7. Metal implants, intracranial surgical clips or pacemakers
8. Weight >450 lbs due to limits for MRI and CT.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents and young adults 13-25 years old with obesity undergoing RYGB or VSG and non-surgical controls.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2015-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Baseline to 24 months change in total and trabecular volumetric BMD (vBMD) (distal radius and tibia) | 2 years

SECONDARY OUTCOMES:
Baseline to 24 month change in bone turnover markers (P1NP and CTX) | 2 years
Baseline to 24 month change in estimated strength measures (FEA of distal radius and tibia) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Madhu Misra, MD, MPH, Principal Investigator — Massachusetts General Hospital; Miriam Bredella, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Tuli S, Lopez Lopez AP, Nimmala S, Pedreira CC, Singhal V, Bredella MA, Misra M. Two-Year Study on the Impact of Sleeve Gastrectomy on Depressive and Anxiety Symptoms in Adolescents and Young Adults with Moderate to Severe Obesity. Obes Surg. 2024 Feb;34(2):568-575. doi: 10.1007/s11695-023-07025-z. Epub 2024 Jan 4. PMID 38177554
- [Derived] Mitchell DM, Singhal V, Nimmala S, Lauze M, Bouxsein ML, Misra M, Bredella MA. Risk of wrist fracture, estimated by the load-to-strength ratio, declines following sleeve gastrectomy in adolescents and young adults. Osteoporos Int. 2024 Feb;35(2):285-291. doi: 10.1007/s00198-023-06941-1. Epub 2023 Oct 21. PMID 37864596
- [Derived] Kaur S, Nimmala S, Singhal V, Mitchell DM, Pedreira CC, Lauze M, Lee H, Stanford FC, Bouxsein ML, Bredella MA, Misra M. Bone changes post-sleeve gastrectomy in relation to body mass and hormonal changes. Eur J Endocrinol. 2023 Sep 1;189(3):346-354. doi: 10.1093/ejendo/lvad121. PMID 37633255
- [Derived] Kaur S, Bredella MA, Misra M, Singhal V. Trajectory of Gonadal Hormones in Adolescent Males up to 2 Years After Sleeve Gastrectomy. Obes Surg. 2023 Oct;33(10):3323-3326. doi: 10.1007/s11695-023-06759-0. Epub 2023 Aug 10. PMID 37561269
- [Derived] Lopez Lopez AP, Tuli S, Lauze M, Becetti I, Pedreira CC, Huber FA, Omeroglu E, Singhal V, Misra M, Bredella MA. Changes in Hepatic Fat Content by CT 1 Year After Sleeve Gastrectomy in Adolescents and Young Adults With Obesity. J Clin Endocrinol Metab. 2023 Nov 17;108(12):e1489-e1495. doi: 10.1210/clinem/dgad390. PMID 37403207
- [Derived] Huber FA, Singhal V, Tuli S, Becetti I, Lopez Lopez AP, Bouxsein ML, Misra M, Bredella MA. Two-year Skeletal Effects of Sleeve Gastrectomy in Adolescents with Obesity Assessed with Quantitative CT and MR Spectroscopy. Radiology. 2023 Jun;307(5):e223256. doi: 10.1148/radiol.223256. PMID 37310246
- [Derived] Mitchell DM, Singhal V, Animashaun A, Bose A, Carmine B, Stanford FC, Inge TH, Kelsey MM, Lee H, Bouxsein ML, Yu EW, Bredella MA, Misra M. Skeletal Effects of Sleeve Gastrectomy in Adolescents and Young Adults: A 2-Year Longitudinal Study. J Clin Endocrinol Metab. 2023 Mar 10;108(4):847-857. doi: 10.1210/clinem/dgac634. PMID 36314507
- [Derived] Nimmala S, Kaur S, Singhal V, Mitchell DM, Stanford FC, Bouxsein ML, Lauze M, Huynh C, Pedreira CC, Lee H, Bredella MA, Misra M. Changes in Sex Steroids and Enteric Peptides After Sleeve Gastrectomy in Youth in Relation to Changes in Bone Parameters. J Clin Endocrinol Metab. 2022 Aug 18;107(9):e3747-e3758. doi: 10.1210/clinem/dgac361. PMID 35689793